CLINICAL TRIAL: NCT00801814
Title: Effect of Adding Escalating Doses of a Novel Highly Viscous Polysaccharide to Either a Liquid or a Solid Test Meal on Post Prandial Glycemia in Healthy Subjects: Determination of the Glycemic Reduction Index Potential (GRIP)
Brief Title: Effect of Escalating Doses of a Novel Viscous Polysaccharide on Postprandial Glycemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Glycemic Index Laboratories, Inc (Industry)
Collaborators: InovoBiologic Inc. (Industry); Canadian Center for Functional Medicine (Other)
Responsible Party: Dr. Alexandra Jenkins, PhD, RD/ Vice President, Glycemic Index Laboratories, Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GIL-5051
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Blood Glucose, Postprandial
Keywords: viscous; fibre; polysaccharide; blood glucose; post prandial
MeSH Terms: interventions — PolyGlycoplex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Placebo Comparator): White Bread
  Interventions: Dietary Supplement: Control
- 2 (Placebo Comparator): White Bread and Margarine Control
  Interventions: Dietary Supplement: Second Control
- 3 (Placebo Comparator): Glucose drink control
  Interventions: Dietary Supplement: Control
- 4 (Experimental): White bread and margarine
  or
  Glucose drink
  Interventions: Dietary Supplement: PolyGlycopleX (PGX); Dietary Supplement: PolyGlycopleX (PG); Dietary Supplement: PolyGlycopleX
- 5 (Experimental): White bread and margarine
  or
  Glucose drink
  Interventions: Dietary Supplement: PolyGlycopleX (PGX); Dietary Supplement: PolyGlycopleX (PG); Dietary Supplement: PolyGlycopleX
- 6 (Experimental): White bread and margarine
  or
  Glucose drink
  Interventions: Dietary Supplement: PolyGlycopleX (PGX); Dietary Supplement: PolyGlycopleX (PG); Dietary Supplement: PolyGlycopleX

INTERVENTIONS:
Dietary Supplement: PolyGlycopleX (PGX) — 2.5 grams of PGX
  Arms: 4; 5; 6
Dietary Supplement: PolyGlycopleX (PG) — 5.0 grams of PGX
  Arms: 4; 5; 6
Dietary Supplement: PolyGlycopleX — 7.5 grams of PGX
  Arms: 4; 5; 6
Dietary Supplement: Control — 0g of PGX
  Arms: 1; 3
Dietary Supplement: Second Control — 0g of PGX
  Arms: 2

SUMMARY:
To determine palatability and extent to which escalating doses of a novel highly viscous polysaccharide [NVP] reduces postprandial glycemia when added to a liquid and a solid meal.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* 18-75 years old
* BMI less than 35 kg/m2

Exclusion Criteria:

* Medications influencing gastrointestinal function
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2006-05 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
postprandial glycemia | Acute study measuring postprandial glucose levels over 2 hours

SECONDARY OUTCOMES:
The glucose reduction index potential (GRIP). The GRIP factor is the reduction in glycemic index units per gram of fiber. | Data analysis

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra L Jenkins, PhD, RD, Study Director — Glycemic Index Laboratories, Inc; Thomas MS Wolever, MD, Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- Glycemic Index Laboratories, Inc., Toronto, Ontario, Canada